CLINICAL TRIAL: NCT00559000
Title: The Efficacy of KIDNET in the Treatment of Traumatized Refugee Children in Germany
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: European Refugee Fund (Other); German Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mb
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: PTSD
Keywords: PTSD; Children; trauma-focused Treatment; KIDNET; Narrative Exposure Therapy for Children
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waitinglist Control (No Intervention)
- KIDNET (Experimental)
  Interventions: Behavioral: KIDNET

INTERVENTIONS:
Behavioral: KIDNET — Narrative Exposure Therapy for Children
  Arms: KIDNET

SUMMARY:
The purpose of the study is to assess the effectiveness of KIDNET in treating traumatized refugee children in Germany

ELIGIBILITY:
Inclusion Criteria:

* refugee children
* age range: 7-16
* PTSD-Diagnosis

Exclusion Criteria:

* none

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2003-12; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
PTSD-Symptoms according to the UCLA Child PTSD INDEX | 1-month, 6-months, 12-months

SECONDARY OUTCOMES:
Cognitive Performance according to SPM, CPM, Rey-Figure-Test, d2; Other mental health disorders according to M.I.N.I.-KID | 6-months, 12-months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Elbert, Prof. Dr., Principal Investigator — University of Konstanz; Martina Ruf, Dipl.-Psych., Principal Investigator — University of Konstanz
Locations (1):
- University of Konstanz, Research and Outpatient Clinic for Refugees, Reichenau-Lindenbühl, Germany

REFERENCES:
- See also: Related Info — http://www.vivo.org